CLINICAL TRIAL: NCT06160011
Title: Effectiveness of Electrical Dry Needdling on Epicondylar Muscle Activation by EMG in Tennis Players. Randomized Clinical Trial
Brief Title: Epicondylar Muscle Activation in Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMGepicondíleos
Record Dates: First submitted 2023-11-20; First posted 2023-12-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Epicondylitis, Lateral
Keywords: Electrical dry needling; EMG; Tennis; Physiotherapy
MeSH Terms: conditions — Tennis Elbow | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group Electrical Dry Needling amd Physiotherapy (Experimental): The intervention group will receive a treatment composed by electrical dry needling and conventional physiotherapy treatment
  Interventions: Other: Electrical dry needling + Conventional physiotherapy
- Intervention Group Dry Needling amd Physiotherapy (Active Comparator): This group will receive a treatment composed by dry needling and conventional physiotherapy treatment
  Interventions: Other: Dry needling + Conventional physiotherapy
- Control Group (Placebo Comparator): Control group will receive conventional physiotherapy treatment
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Electrical dry needling + Conventional physiotherapy — Electrical dry needling and conventional physiotherapy treatment (massage, pressure release): 2 sessions
  Arms: Intervention Group Electrical Dry Needling amd Physiotherapy
Other: Dry needling + Conventional physiotherapy — Dry needling and conventional physiotherapy treatment (massage, pressure release): 2 sessions
  Arms: Intervention Group Dry Needling amd Physiotherapy
Other: Conventional physiotherapy — Conventional physiotherapy treatment (massage, pressure release): 2 sessions
  Arms: Control Group

SUMMARY:
Epicondylitis is one of the most common pathologies in tennis players. The search for an effective treatment is necessary for the relief of symptoms and the return to sports practice. Therefore, a ddry needling treatment in combination with electricity is postulated as an alternative to isolated dry needling treatment or conventional physiotherapy treatment. Data will be collected in relation to pain and muscle activation by EMG in order to check the effectiveness of these techniques as well as the muscle activation that is generated.

ELIGIBILITY:
Inclusion Criteria:

* tennis players of both sexes
* federated and non-federated of Castilla y León
* playing tennis for at least 2 years
* presence if one trigger point in epicondilar musculature

Exclusion Criteria:

* not informed consent signature
* nervous, vascular, articular or musculoskeletal system alterations
* tests or techniques performed fear (belonephobia)
* pregnancy
* allergic to any type of metal or body oil
* active febrile proces
* current pain treatments in the area involved
* surgery in the last year for upper limb pathologies
* cognitive alterations
* taking painkillers or anti-inflammatory drugs 24 hours before the start of the study or taking them during the duration of the study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Muscular activation | 30 minutes
  Electromyography: the adequate electrical activity of the muscles will be observed and the nerves will show adequate conduction of electrical impulses. This indicates normal and healthy functioning of the neuromuscular system
Subjective Pain | Initial, up to 2 weeks, and up to 6 weeks
  Numeric Pain Rating Scale: Single 11-point numerical scale where scores correspond to Pain scores are interpreted as: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain and 7-10 = severe pain. 7-10 = severe pain
Algometry | Initial, up to 2 weeks, and up to 6 weeks
  Pressure algometer is an instrument with a circular disk on which the pressure measurements are displayed (with a range of 5 kg, divided into 10 parts of half a kilogram), and a rubber tip with a circular surface of 1 cm2, which allows transferring the pressure force to deep tissues.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No